CLINICAL TRIAL: NCT04521452
Title: An Open-label, Randomized Study of Inhibitory Effect of Evogliptin, the Dipeptidyl Peptidase-4 Inhibitor, on the Progression of Aortic Valve Calcification in Patients With Type 2 Diabetes Mellitus and Mild-to-moderate Aortic Stenosis
Brief Title: Randomized, Open-label Trial of Inhibitory Effect of Evogliptin on Progression of CAVD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: REDNVIA Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jae-Kwan Song, CMO, M.D, Ph.D, FACC, Department of Cardiology, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIP_CAVD_DM
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: CAVD
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Intervention Model Description: Randomized, open-label trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evogliptin Group (Experimental): evogliptin 5mg daily
  Interventions: Drug: Evogliptin
- Non-evogliptin Group (No Intervention): DM medications except evogliptin and other DPP-4 inhibitors

INTERVENTIONS:
Drug: Evogliptin — Subjects will receive evogliptin 5 mg daily
  Arms: Evogliptin Group

SUMMARY:
The purpose of this study is to assess an inhibitory effect of Evogliptin on the progression of mild-to-moderate aortic stenosis in patients with T2DM and calcific aortic stenosis.

DETAILED DESCRIPTION:
Despite a lot of clinician's efforts to develop an effective medical treatment of calcific aortic valve disease (CAVD) for decades, there is no scientifically-proved medical treatment yet. Since the pathological features of CAVD are characterized by inflammatory cell infiltration and lipid deposition, as in atherosclerosis, statin drugs that are proved to be effective in the treatment of cardiovascular disease, have been used in the most recent randomized clinical trials; however, different types of medications showed negative results and thus, CAVD represents an unmet clinical need.

Researchers of Asan Medical Center have proved that dipeptidyl-peptidase-4 (DPP-4)-IGF (insulin-like growth factor)-1 axis is important for pathologic osteoblast transformation of valvular interstitial cell (VIC), and reported that the administration of DPP-4 inhibitor prevents the calcification effectively in the actual animal model of CAVD. Under a normal condition, IGF-1 suppresses the pathologic transformation of VIC; however, when endothelial cells are damaged due to aging or various pathological conditions, DPP-4 expression is increased in valvular tissue. Since DPP-4 acts as an enzyme that degrades IGF-1, it reduces normal IGF-1 activity and increases transformation of VIC to osteoblast, causing pathological calcification and worsening CAVD.

After comparing six different DPP-4 inhibitors, researchers of Asan Medical Center discovered that evogliptin has higher cardiac tissue distribution compared to other DPP-4 inhibitors. In addition, the DPP-4 inhibitors with high cardiac tissue distribution have shown decreased incidence rate of severe CAVD in the retrospective study. Based on these findings, this study will examine the effect of evogliptin on progression of CAVD.

The study is a randomized, open-label trial of evogliptin in subjects with T2DM and moderate-to-severe CAVD. Subjects who have agreed to participate in the study and signed the ICF will undergo a screening period and those who meet the eligibility criteria will be randomized in a 1:1 ratio to evogliptin or non-evogliptin group. The subjects will take the drug for 96 weeks and will be closely monitored for efficacy. The effectiveness of evogliptin on inhibition of CAVD progression will be evaluated by comparing the change in aortic valve calcium volume in the evogliptin group against that of the non-evogliptin group.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 19 years or older
2. Subjects who were diagnosed with type 2 diabetes mellitus and being treated with oral hypoglycemic drugs
3. Subjects whose Doppler echocardiography or Heart CT performed within 8 weeks prior to or during Screening Visit (Visit 1) is satisfying any of the followings:

   * Doppler echocardiogrphy (aortic valve calcification and/or hypertrophy with aortic peak velocity≥2.0 m/s); or
   * Heart CT (aortic valve calcium score≥300 AU)
4. Subjects who decided to take part in this study on his/her own volition after listening to the details of this study

Exclusion Criteria:

1. Subjects with severe aortic valve stenosis (aortic peak velocity>4.0 m/s, mean pressure gradient >40 mmHg, or aortic valve area≤0.75 cm2)
2. Subjects with left ventricular ejection fraction < 40%
3. Heart failure patients: Subjects with heart failure of NYHA functional class II-IV
4. Subjects with an estimated glomerular filtration rate (eGFR) of <30ml
5. Subjects with type 1 diabetes or diabetic ketoacidosis
6. Subjects with serious hypersensitivity to DPP-4 inhibitors
7. Subjects who have received/are receiving any of the following medication therapies:

   * Vitamin K
   * Calcium supplement (or osteoporosis medication)
8. Subjects whose aortic valve stenosis is not caused by degenerative or bicuspid valve disease (e.g. rheumatic valve disease)
9. Subjects who have received or are expected to receive (as of Visit 1) aortic valve surgery during the study.
10. Subjects for whom a two-year clinical course investigation is not possible due to malignant tumor or cerebrovascular disease
11. Pregnant or lactating women
12. Women of childbearing potential who are sexually active and do not agree to use proper contraception during the study

    * Proper contraception means physical barrier method including condom, contraceptive diaphragm or cervix cap. The use of contraceptive or oral contraceptive containing hormones that may induce drug-drug interaction with the investigational product is not allowed during the study (with the exception of an oral contraceptive administered to cure menopausal symptoms, only if the dosage has been consistent for the past 8 weeks)
13. Any other subjects deemed not eligible for this study by an investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in aortic valve calcium volume at week 96 from baseline | 96 weeks

SECONDARY OUTCOMES:
Change in aortic valve calcium volume at week 48 from baseline | 96 weeks
Change in aortic valve calcium score at week 48 and week 96 from baseline | 48 weeks, 96 weeks
Rate of change (%) in aortic valve calcium volume at week 48 and week 96 from baseline | 48 weeks, 96 weeks
Change in peak aortic-jet velocity at week 48 and week 96 from baseline | 48 weeks, 96 weeks
Change in aortic peak & mean pressure gradient at week 48 and week 96 from baseline | 48 weeks, 96 weeks
Change in aortic valve area at week 48 and week 96 from baseline | 48 weeks, 96 weeks
Time of major cardiovascular event | anytime during the entire follow-up of 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Lindman BR, Clavel MA, Mathieu P, Iung B, Lancellotti P, Otto CM, Pibarot P. Calcific aortic stenosis. Nat Rev Dis Primers. 2016 Mar 3;2:16006. doi: 10.1038/nrdp.2016.6. PMID 27188578
- [Background] Bonow RO, Greenland P. Population-wide trends in aortic stenosis incidence and outcomes. Circulation. 2015 Mar 17;131(11):969-71. doi: 10.1161/CIRCULATIONAHA.115.014846. Epub 2015 Feb 17. No abstract available. PMID 25691712
- [Background] Choi B, Lee S, Kim SM, Lee EJ, Lee SR, Kim DH, Jang JY, Kang SW, Lee KU, Chang EJ, Song JK. Dipeptidyl Peptidase-4 Induces Aortic Valve Calcification by Inhibiting Insulin-Like Growth Factor-1 Signaling in Valvular Interstitial Cells. Circulation. 2017 May 16;135(20):1935-1950. doi: 10.1161/CIRCULATIONAHA.116.024270. Epub 2017 Feb 8. PMID 28179397
- [Background] Otto CM, Lind BK, Kitzman DW, Gersh BJ, Siscovick DS. Association of aortic-valve sclerosis with cardiovascular mortality and morbidity in the elderly. N Engl J Med. 1999 Jul 15;341(3):142-7. doi: 10.1056/NEJM199907153410302. PMID 10403851
- [Background] Aronow WS, Ahn C, Shirani J, Kronzon I. Comparison of frequency of new coronary events in older subjects with and without valvular aortic sclerosis. Am J Cardiol. 1999 Feb 15;83(4):599-600, A8. doi: 10.1016/s0002-9149(98)00922-9. PMID 10073870
- [Background] Pawade TA, Newby DE, Dweck MR. Calcification in Aortic Stenosis: The Skeleton Key. J Am Coll Cardiol. 2015 Aug 4;66(5):561-77. doi: 10.1016/j.jacc.2015.05.066. PMID 26227196
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Brandenburg VM, Reinartz S, Kaesler N, Kruger T, Dirrichs T, Kramann R, Peeters F, Floege J, Keszei A, Marx N, Schurgers LJ, Koos R. Slower Progress of Aortic Valve Calcification With Vitamin K Supplementation: Results From a Prospective Interventional Proof-of-Concept Study. Circulation. 2017 May 23;135(21):2081-2083. doi: 10.1161/CIRCULATIONAHA.116.027011. No abstract available. PMID 28533322